CLINICAL TRIAL: NCT05254184
Title: Pooled Mutant KRAS-Targeted Long Peptide Vaccine Combined With Nivolumab and Ipilimumab for Patients With Advanced KRAS Mutated Non-Small Cell Lung Cancer
Brief Title: KRAS-Targeted Vaccine With Nivolumab and Ipilimumab for Patients With NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J21131; IRB00306311 (Other: Johns Hopkins University SOM)
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Advanced KRAS mutated Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients With NSCLC (Experimental): All participants will receive the intervention.
  Interventions: Drug: Pooled Mutant KRAS-Targeted Long Peptide Vaccine 0.3mg each; 1.8mg total peptides

INTERVENTIONS:
Drug: Pooled Mutant KRAS-Targeted Long Peptide Vaccine 0.3mg each; 1.8mg total peptides — administering the KRAS peptide vaccine with poly-ICLC adjuvant in combination with nivolumab and ipilimumab
  Other Names: Nivolumab 3 mg/kg every 2 weeks; Ipilimumab 1 mg/kg every 6 weeks

SUMMARY:
This is a single institution, Phase 1 study for patients with Stage III/IV unresectable Kirsten rat sarcoma (KRAS) mutated NSCLC to evaluate safety of the pooled mutant-KRAS peptide vaccine (KRAS peptide vaccine) with polyinosinic-polycytidylic acid (poly-ICLC) adjuvant in combination with nivolumab and ipilimumab in the first line treatment setting. The primary objectives of this study are to determine the safety and feasibility of administering the KRAS peptide vaccine with poly-ICLC adjuvant in combination with nivolumab and ipilimumab. The secondary objectives are to estimate the progression free survival (PFS) of pooled mutant-KRAS long peptide vaccine with poly-ICLC adjuvant in combination with Ipilimumab + Nivolumab for the first line treatment of patients with unresectable Stage III/IV NSCLC whose tumors harbor selected KRAS mutations (KRAS glycine-to-cysteine substitution at codon 12 (G12C), KRAS glycine-to-valine substitution at codon 12 (G12V), KRAS glycine-to-Detoxglyphosate substitution at codon 12 (G12D), KRAS glycine-to-arginine substitution at codon 12 (G12A), KRAS glycine-to-Aspartic Acid "D" at codon 13 (G13D) or KRAS G12R) and to assess the impact of predicted KRAS mutations on mutant-KRAS specific T cell responses in the peripheral blood of these patients. Exploratory objectives will assess the impact of predicted KRAS mutations on mutant-KRAS specific T cell responses in the peripheral blood, as well as changes in circulating tumor deoxyribonucleic acid (ctDNA). Approximately 15 subjects will be enrolled to have 12 evaluable subjects for T cell response assessment. Safety analysis will include all enrolled patients who receive at least one dose of vaccine. The evaluable population for T cell response will consist of all patients who receive at least one dose of vaccine and have baseline and post-treatment T cell measures in the peripheral blood at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-proven adenocarcinoma of the lung deemed to be locally advanced/unresectable or metastatic as per American Joint Committee on Cancer (AJCC) version 8, who has not received prior therapy for this stage of disease.

  • Prior therapy for early stage NSCLC allowed. Progressive disease after at least 6 months of anti-programmed death (PD) ligand therapy (anti-PD-L1 therapy) (i.e. Durvalumab) for Stage III disease is allowed.
* Must have tumor lesions amenable to repeated biopsy, and patient's acceptance to have a tumor biopsy of an accessible lesion at baseline and on treatment if the lesion can be biopsied with acceptable clinical risk (as judged by the Principal Investigator).
* Measurable disease as defined by RECIST v1.1.
* Have one of the six KRAS mutations (KRAS G12C, KRAS G12V, KRAS G12D, KRAS G12A, KRAS G13D or KRAS G12R) in vaccine expressed in tumor as defined by a Clinical Laboratory Improvement Amendments (CLIA) certified tumor or plasma based genomic testing platform performed either through a local laboratory or through the investigators' central laboratory.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Appendix A).
* Patients must have adequate organ and marrow function as defined below:

Microliters (mcL) Microliter (uL)

* Leukocytes ≥ 3,000/mcL
* Lymphocytes > 500/mm3
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 75 × 103/uL
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 1.5 x ULN (< 2.0 x ULN for subjects with documented Gilbert's syndrome)
* aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT)(SGPT)≤ 2.5 × ULN (if liver metastases are present, ≤ 5 x ULN)
* Alkaline phosphatase ≤5.0 × ULN
* Creatinine ≤1.5 × ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 0.85 / 72 x serum creatinine in mg/dL

Male CrCl = (140 - age in years) x weight in kg x 1.00 / 72 x serum creatinine in mg/dL

* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG). WOCBP is defined in Section 4.6. Note: If a patient has a positive or indeterminate serum or urine pregnancy test, then an ultrasound must be done to rule out pregnancy to enroll on trial.
* WOCBP must agree to follow instructions for method(s) of contraception from the time of enrollment for the duration of treatment with study drug(s) plus 5 half-lives of study drug(s) plus 4 weeks (duration of ovulatory cycle) for a total of 5 months post treatment completion.
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug(s) plus 90 days (duration of sperm turnover) for a total of 7 months post-treatment completion.
* At least one barrier method of contraception must be employed by all sexually active patients (male and female), regardless of other methods, to prevent the transfer of body fluids.
* Ability to understand and willingness to sign a written informed consent document.
* Last dose of adjuvant chemotherapy or radiation therapy administered within 6 months of screening date

Exclusion Criteria:

* Patient is expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Any of the following procedures or medications:
* Within 2 weeks prior to initiation of study treatment:

  * Systemic or topical corticosteroids at immunosuppressive doses (> 10 mg/day of prednisone or equivalent). Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
  * Palliative or adjuvant radiation or gamma knife radiosurgery.
  * Chemotherapy
* Within 4 weeks prior to initiation of study treatment:

  * Any investigational cytotoxic drug. Exposure to any cytotoxic drug within 4 weeks or 5 half-lives (whichever is shorter) is prohibited. If 5 half-lives are shorter than 4 weeks, agreement with Investigational New Drug (IND) Sponsor is mandatory.
  * Any investigational device
  * Non-oncology vaccines containing live virus. Examples include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Influenza, pneumonia vaccines (polysaccharide and conjugated forms) and Corona Virus Disease 2019 (COVID-19) vaccines will be allowed, however the investigators recommend that subjects not receive any dose of vaccine within 7 days before or after the subjects' scheduled KRAS peptide vaccination.
  * Allergen hyposensitization therapy.
  * Growth factors, e.g. granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin
  * Major surgery (excludes celiac plexus block, biliary stent placement, and other minor procedures such as dental work, skin biopsy, etc.).
* Patients with a history of prior treatment with immunotherapy agents (including, but not limited to: Interleukin 2 (IL-2), interferon, anti-PD-L2, anti-cluster of differentiation 137 (anti-CD137), anti-oxidation (OX) 40 (anti-OX-40), anti-cluster of differentiation 40 (anti-CD40), anti-cytotoxic T-lymphocyte-associated (CTLA) antigen 4 (anti-CTLA-4), or anti-lymphocyte activating gene (LAG) 3 (anti-LAG-3) antibodies).

  * Prior anti-PD-(L)1 therapy for non-metastatic NSCLC (ie/Durvalumab) is allowed if patient had received at least 6 months of therapy prior to having disease progression.
* History of severe hypersensitivity reaction to any monoclonal antibodies or related compounds or to any of these agents' components (e.g., history of severe hypersensitivity reactions to drugs formulated with polysorbate 80).

  * This includes any prior immunotherapy agents; patients having toxicity with prior anti-PD-L1 therapy requiring cessation of treatment must be excluded.
* Untreated or symptomatic brain metastases.

  * Treated brain metastases allowed on study if asymptomatic and therapy was completed at least 2 weeks prior to treatment start, and steroid dosing is as 3.2.2
* Has an active known or suspected autoimmune disease or which has required systemic therapy in the last 2 years. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Known history of interstitial lung disease or of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a pulse oximetry < 90% on room air.
* Requires the use of home oxygen.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV1/2 antibodies), hepatitis B, or hepatitis C infection.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness that would limit compliance with study requirements.
* Patients who have been diagnosed with another cancer or myeloproliferative disorder in the past 5 years except for superficial bladder cancer, non-melanoma skin cancers, or a low grade prostate cancer not requiring therapy.
* Has a diagnosis of immunodeficiency.
* Presence of any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft. Patients with a history of allogeneic hematopoietic stem cell transplant will be excluded.
* Any other sound medical or psychiatric reason as determined by the Investigator.
* Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or other substance abuse (including alcohol) that could potentially interfere with adherence to study procedures or requirements.
* Patient is unwilling or unable to follow the study schedule for any reason.
* Patient is pregnant or breastfeeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety of administering a KRAS peptide vaccine in combination with nivolumab and ipilimumab as assessed by adverse events | Up to day 29
  The safety of administering a KRAS peptide vaccine in combination with nivolumab and ipilimumab will be assessed by the occurrence of the following adverse events:
  * Grade 3 or above drug-related toxicities
  * Drug-related toxicity by grade
  * Vaccine site reactions after KRAS injections
  * Nivolumab-related infusion reactions
  * Ipilimumab-related infusion reactions
  * Immune-related adverse events (AEs)
  * Unacceptable toxicities
  * Treatment-emergent changes from normal to abnormal values in key laboratory parameters
Feasibility of administering a KRAS peptide vaccine in combination with nivolumab and ipilimumab as assessed by adverse events | Up to 29 days
  Feasibility of administering a KRAS peptide vaccine in combination with nivolumab and ipilimumab will be assessed by the occurrence of the following adverse events:
  * Grade 3 or above drug-related toxicities
  * Drug-related toxicity by grade
  * Vaccine site reactions after KRAS injections
  * Nivolumab-related infusion reactions
  * Ipilimumab-related infusion reactions
  * Immune-related adverse events (AEs)
  * Unacceptable toxicities
  * Treatment-emergent changes from normal to abnormal values in key laboratory parameters

SECONDARY OUTCOMES:
Progression Free Survival (PFS) as assessed by imaging | Baseline to progression, up to 4 years
  PFS as defined as the time from first vaccination to the earliest evidence of progressive disease (based on imaging) or death from any cause as determined by medical history and physical examination in combination with imaging evaluation, cytology, or tissue biopsy.
Change in interferon-producing mutant-KRAS-specific cluster of differentiation (CD) 8 T cells in the peripheral blood | Pre-vaccination baseline to end of treatment, up to 2 years
  T cell response will be evaluated by the fold change in interferon-producing mutant-KRAS-specific CD 8 T cells in the peripheral blood.
Change in interferon-producing mutant-KRAS-specific CD 4 T cells in the peripheral blood | Pre-vaccination baseline to end of treatment, up to 2 years
  T cell response will be evaluated by the fold change in interferon-producing mutant-KRAS-specific CD 4 T cells in the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Marrone, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No